CLINICAL TRIAL: NCT03721874
Title: MaasFlex: Double-Blind, Randomized, Phase IV, Mechanistic, Placebo-Controlled, Cross-Over, Single-Center Study to Evaluate the Effects of 2 Weeks Dapagliflozin Treatment on Nocturnal Substrate Oxidation, Glucose Metabolism and Muscle Mitochondrial Function in Individuals With Impaired Glucose Homeostasis
Brief Title: Effects of 2 Weeks Treatment With Dapagliflozin in Subjects With an Impaired Glucose Homeostasis on Nocturnal Substrate Oxidation
Acronym: MaasFlex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Patrick Schrauwen, Prof. Dr., Maastricht University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL67170.068.18
Record Dates: First submitted 2018-10-23; First posted 2018-10-26 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Prediabetic State; Substrate Oxidation
Keywords: Dapagliflozin; Disrupted glucose homeostasis; Nocturnal substrate oxidation; Glucose metabolism
MeSH Terms: conditions — Prediabetic State | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Double-Blind, Randomized, Phase IV, Mechanistic, Placebo-Controlled, Cross-Over, Single-Center Study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin 10 mg (Active Comparator): Patients will receive dapagliflozin 10 mg in tablet for a maximum of 14 days based on randomization sequence in Period 1.
  Patients that received 10 mg dapagliflozin in the first treatment period will receive matching placebo in the second treatment period for a maximum of 14 days.
  Interventions: Drug: Dapagliflozin 10mg
- Placebo matching to dapagliflozin 10 mg (Placebo Comparator): Patients will receive matching placebo in tablet for a maximum of 14 days based on randomization sequence.
  Patients who received placebo in the first treatment will receive 10 mg dapagliflozin in the second treatment period, for a maximum of 14 days
  Interventions: Drug: Placebo matching to Dapagliflozin 10 mg

INTERVENTIONS:
Drug: Dapagliflozin 10mg — The study consist of 2 weeks treatment period 1, 6-8 weeks wash-out period and 2 weeks treatment period 2.
  The subject may be administered dapagliflozin 10 mg during Period 1 or Period 2.
  Arms: Dapagliflozin 10 mg
Drug: Placebo matching to Dapagliflozin 10 mg — The study consist of 2 weeks treatment period 1, 6-8 weeks wash-out period and 2 weeks treatment period 2.
  The subject may be administered placebo during Period 1 or Period 2.
  Arms: Placebo matching to dapagliflozin 10 mg

SUMMARY:
The purpose of this study is to investigate the effect of 2 weeks dapagliflozin treatment in individuals with a disrupted glucose homeostasis on the switch between carbohydrate and lipid oxidation during the night

DETAILED DESCRIPTION:
To investigate if dapagliflozin improves nocturnal substrate oxidation expressed as respiration quotient (RQ) during the sleeping period in comparison with placebo after 2-weeks double blind treatment in subjects with a disrupted glucose homeostasis.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent prior to any study specific procedures.
2. Males aged ≥ 40 and ≤ 75 years and post-menopausal women (defined as at least 1 year post cessation of menses) aged ≥ 50 and ≤ 75 years
3. Body mass index (BMI) ≥ 27 and ≤ 38 kg/m2.
4. Sedentary lifestyle (not more than 3 hours of programmed exercise per week).
5. Stable dietary habits.
6. Impaired glucose homeostasis based on one or a combination of the following criteria:

   * Impaired Glucose Tolerance (IGT): plasma glucose values ≥ 7.8 mmol/l and ≤ 11.1 mmol/l 120 minutes after consumption of the glucose drink during the 2h, 3-point OGTT.
   * Impaired Fasting Glucose (IFG): fasting plasma glucose ≥ 6.1 mmol/l and ≤ 6.9 mmol/l.
   * Insulin Resistance: glucose clearance rate ≤ 360 ml/kg/min, as calculated by Oral Glucose Insulin Sensitivity 120 (OGIS120) model based on the 2h, 3-point OGTT.
   * HbA1c ≥ 5.7% and ≤ 6.4%.

Exclusion Criteria:

1. Clinical diagnosis of Type 1 or 2 Diabetes Mellitus.
2. Active cardiovascular disease: participants who experienced a heart attack in the last year, or participants who are currently under regular control of a physician for a heart condition.
3. Weight gain or loss > 5 kg in the last 3 months, ongoing weight-loss diet (hypocaloric diet) or use of weight loss agents.
4. Regular smoking and other regular nicotine use.
5. Anaemia.
6. Uncontrolled hypertension.
7. Clinically significant out of range values of serum levels of either alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) in the Investigator's opinion.
8. Unstable or rapidly progressing renal disease or estimated Glomerular Filtration Rate (eGFR) <60 mL/min (Cockcroft-Gault formula).
9. Use of anti-coagulant treatment and other concomitant medication will be evaluated on a case to case basis with a general physician.
10. Use of medication such as oral glucocorticoids, anti-estrogens or other medications that are known to markedly influence insulin sensitivity.
11. Use of loop diuretics.
12. Intake of dietary supplements except multi-vitamins and minerals.
13. Alcohol consumption of > 14 drinks per week for women and > 21 drinks per week for men (1 drink = 35 cl beer, 14 cl wine or 4 cl hard liquor).
14. Known hypersensitivity to dapagliflozin or any of the excipients of the product.
15. For women only - currently pregnant (confirmed with positive pregnancy test) or breast-feeding.
16. Participation in another biomedical study within 1 month before the screening visit.
17. Any contraindication for MRI scanning.
18. Participants who do not want to be informed about unexpected medical findings, or do not wish that their physician be informed about coincidental findings, cannot participate in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Change in nightly substrate oxidation measured as respiration quotient (RQ) during the sleeping period | From screening to day 14
  Comparison of dapagliflozin versus placebo after 14 days of treatment on nightly substrate oxidation as measured by respiratory quotient (VCO2/VO2) during the sleeping period.

SECONDARY OUTCOMES:
Change in morning and late afternoon hepatic glycogen content | 1 hour
  Comparison of dapagliflozin versus placebo after 14 days of treatment on hepatic glycogen content determined by non-invasive 13C-MRS (magnetic resonance spectroscopy) in the morning and evening
Change in 24h substrate oxidation as determined by indirect calorimetry in a whole-body respiratory chamber and based on urinary nitrogen excretion | 24 hours
  Comparison of dapagliflozin versus placebo after 14 days of treatment on 24h substrate oxidation as determined by indirect calorimetry in a whole-body respiratory chamber and based on urinary nitrogen excretion
Change in 24h plasma markers | 24 hours
  Comparison of dapagliflozin versus placebo after 14 days of treatment on 24h plasma markers including plasma glucose, NEFA, total amino acid levels incl BCAA levels, insulin and glucagon
Change in muscle mitochondrial function | 60 minutes
  Comparison of dapagliflozin versus placebo after 14 days of treatment on muscle mitochondrial function as determined by high resolution respirometry
Change in intrahepatic lipid content and composition | 45 minutes
  Comparison of dapagliflozin versus placebo after 14 days of treatment on intrahepatic lipid content and composition as determined by non-invasive 1H-MRS (magnetic resonance spectroscopy )
Change in intramyocellular lipid content and composition - including acylcarnitine levels | 45 minutes
  Comparison of dapagliflozin versus placebo after 14 days of treatment on intramyocellular lipid content and composition-including acylcarnitine levels as determined in muscle biopsies
Change in muscle glycogen content | 45 minutes
  Comparison of dapagliflozin versus placebo after 14 days of treatment on muscle glycogen content as determined biochemically in muscle biopsies
Change in systolic and diastolic blood pressure | 45 minutes
  Comparison of dapagliflozin versus placebo after 14 days of treatment on systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, Prof. dr., Principal Investigator — principle investigator
Locations (1):
- Maastricht University and Medical Centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Veelen A, Andriessen C, Op den Kamp Y, Erazo-Tapia E, de Ligt M, Mevenkamp J, Jorgensen JA, Moonen-Kornips E, Schaart G, Esterline R, Havekes B, Oscarsson J, Schrauwen-Hinderling VB, Phielix E, Schrauwen P. Effects of the sodium-glucose cotransporter 2 inhibitor dapagliflozin on substrate metabolism in prediabetic insulin resistant individuals: A randomized, double-blind crossover trial. Metabolism. 2023 Mar;140:155396. doi: 10.1016/j.metabol.2022.155396. Epub 2022 Dec 30. PMID 36592688